CLINICAL TRIAL: NCT01377688
Title: Personalized Diabetic Kidney Disease Risk Info to Initiate and Maintain Health Behavior Changes
Acronym: DKDPilot
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00030501
Record Dates: First submitted 2011-06-20; First posted 2011-06-21 (Estimated); Last update posted 2014-06-03 (Estimated); Status verified 2014-03

CONDITIONS: Diabetic Kidney Disease
Keywords: DKD
MeSH Terms: conditions — Diabetic Nephropathies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Diabetics with PKD: Diagnoses of diabetes type 2 with progressive kidney disease (slope of eGFR decline between -15 to -3 ml/min/1.73m2 per year, estimated by calculating an eGFR for each creatinine using the 4-variable Modification of Diet in Renal Disease Study [MDRD] equation and conducting a simple ordinary least squares regression from these values to evaluate changes over time to derive each individuals' slope of eGFR, annualized using test dates)

SUMMARY:
We propose to pilot a telehealth approach to evaluate components of risk communication by:

1. Providing personalized tailored patient feedback to help initiate and maintain specific diabetic kidney disease (DKD)-related behaviors (e.g., medication adherence, weight, exercise, diet, smoking cessation) to reduce their risks.
2. Evaluating how this feedback can be incorporated into clinical care by examining 6 month patient outcomes.

Specific Aims are:

1. To evaluate the feasibility and acceptability of providing both patients and their provider feedback on individuals' DKD risk via the telehealth intervention and incorporating it into regular clinical practice.
2. If improvements in outcomes are found, to estimate the cost of the program in terms of the patient, provider, and overall costs of implementing the program.

DETAILED DESCRIPTION:
We propose an innovative telehealth approach that has reduced antecedents of kidney disease, including poor blood pressure and glucose control, but has never been used to treat DKD. To mitigate the growing burden of DKD, these studies are designed to determine whether a potentially scalable, telehealth intervention effectively slows progression of DKD in a diverse US population and whether it is also cost-effective. The intervention simultaneously addresses medication management and behavioral therapies and education that seek to optimize adherence and self-efficacy. This proposed pilot trial will begin to evaluate if a multifactorial telehealth intervention may be effective in reducing progression of DKD.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of diabetes with progressive kidney disease

Exclusion Criteria:

* Metastatic cancer
* Dementia
* Psychosis
* No Access to phone
* Diagnosis of non-diabetic kidney disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetics with progressive kidney disease
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2011-10; Primary Completion 2014-04 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Blood pressure and /or Estimated Glomerular Filtration Rate (eGFR) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Hayden B Bosworth, PhD, Principal Investigator — Duke Universtiy Medical Center
Locations (1):
- Duke University Health System, Durham, North Carolina, United States